CLINICAL TRIAL: NCT06537271
Title: Effect of Web-Based Animated Training Given To Mothers With Children Between 18-36 Months on The Awareness Level: Mother-Child School
Brief Title: Web-Based Animated Training:Mother-Child School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Igdir University (Other)
Responsible Party: Principal Investigator, Eda Gulbetekin, Assist. Prof. Principal Investigator, Igdir University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Eda2
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Toilet Training; Autism; Breast Feeding
Keywords: toilet training; autism; weaning ending
MeSH Terms: conditions — Autistic Disorder; Breast Feeding | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Participation in the study is entirely voluntary. After the purpose of the study is explained to the experimental group by the researcher and written and verbal permission is obtained from those who voluntarily agree to participate in the study, the pre-test data will be collected by the researcher.
  Interventions: Combination Product: experimental group
- Control Group (Experimental): After the purpose of the study is explained to the control group by the researcher and written and verbal permission is obtained from those who voluntarily agree to participate in the study, the pre-test data will be collected by the researcher.At the end of 8 weeks, the researcher will fill out the questionnaire forms for the experimental group and collect post-test data.
  Interventions: Combination Product: Control Group

INTERVENTIONS:
Combination Product: experimental group — Autism awareness, breastfeeding cessation and toilet training knowledge and attitude training guide and weekly training content animation videos will be prepared for the experimental group and uploaded via WhatsApp and training will be provided. All participants will be interviewed face to face before the training and the necessary information about our study will be provided. Feedback will be received from the researcher regarding the videos, and participants in the study will be able to ask their questions via WhatsApp and share digital content in a digital environment. Evaluation will be made by conducting group work with individuals. Reminders such as mobile phone messages will be used. Training will be carried out within an 8-week program. Each week, training videos on the topics prepared in line with the training guide will be prepared and shared via WhatsApp. Feedback will be received by creating interactive communication environments.
  Arms: experimental group
Combination Product: Control Group — After the purpose of the study is explained to the control group by the researcher and written and verbal permission is obtained from those who voluntarily agree to participate in the study, the pre-test data will be collected by the researcher.At the end of the training, survey forms will be filled out by the researcher for the control group and post-test data will be collected.
  Arms: Control Group

SUMMARY:
Introduction: Toilet training is the training that helps children gain control of their urine and stool while they are asleep and awake, and to recognize that they need to go to the toilet and relieve themselves without being reminded or helped.Toilet training is the training that helps children gain control of their urine and stool while they are asleep and awake, and to recognize that they need to go to the toilet and relieve themselves without being reminded or helped.Weaning is the gradual cessation of breastfeeding. For most mothers and their babies, weaning can be a very difficult situation. It is extremely important to support breastfeeding and to wean at a time that is convenient for the mother and baby.

Purpose: This study aims to examine the effects of web-based animation-based education given to mothers with children aged 18-36 months on the level of awareness.

Material Method:The research was planned as an experimental study with experimental and control groups.In collecting the data, "Personal Information Form", "Toilet Training Knowledge and Attitude Scale", "Autism Awareness Scale Mother Form", "Breastfeeding Termination Scale" and "Informed Voluntary Consent Form" will be used.The universe of the study will consist of parents with children between 18-36 months of age. The sample of the study was calculated using the GPower computer program. With the power analysis, it was found that a total of 70 patients should be included in the control group and the experimental group, 35 patients each, in the calculation made at the α = 0.05 error level, the effect size for large independent groups, d = 0.8 for the t test and 95% power of the study.

DETAILED DESCRIPTION:
Toilet training is a developmental task that affects families with young children, which occurs when the child develops the ability to urinate and defecate at the appropriate time and environment. Toilet training begins when the child becomes aware of his/her limits and learns to control his/her behavior and instinctive impulses. Parents' approaches and social expectations should be parallel to developmental periods. This is necessary for the child to realize himself/herself.

Mothers may need training due to their inadequate knowledge and attitudes about starting and continuing toilet training. Nurses play an important role in preventing parents' incorrect toilet training knowledge and attitudes in this regard.

Autism spectrum disorder (ASD), also known as autism, is a common, highly hereditary and heterogeneous neurodevelopmental disorder that has underlying cognitive characteristics and usually occurs together with additional health problems.

Autism is usually associated with poor emotional control, anxiety and impulsivity. Challenging behaviors, including aggression towards others, are observed in autistic individuals and are not socially accepted. Increasing awareness about autism will allow the differences of autistic individuals to be understood and the correct approach to be provided in social areas. Researching autism awareness in children during this period is important so that mothers can both observe their own children better and raise awareness about their children's approach to their friends.

Weaning is the gradual termination of breastfeeding. The breastfeeding period is a special process in which the bond of love between most mothers and their babies is established, strengthened and developed. During this period, it can be quite difficult for most mothers and their babies to end breastfeeding. The sudden end of this process, which is a joy for the baby, can cause problems in the emotional, social and cognitive development of the child in the future.

It is extremely important to support breastfeeding and to end breastfeeding at a time that is suitable for the mother and the baby with the right method.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to Participate in the Study
* Parents with children between 18-36 months of age who agree to participate in the study
* Being literate in Turkish
* Having a computer or mobile phone and internet connection at home
* Being able to use Whatsapp
* Not having a visual or auditory health problem that would prevent participation in the study
* Not having a communication barrier

Exclusion Criteria:

* Having a visual or auditory health problem that would prevent participation in the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Autism Awareness Scale of Mothers of Preschool Children | for 8 weeks, once a week
  It consists of 23 questions on a 4-point Likert type (1=False, 2=Undecided, 3=Partially True, 4=Absolutely True). Possible scores range from 23 to 92. An increase in the total score indicates a higher level of awareness. Cronbach's alpha value was 0.947 and it was determined that it had a two-factor structure (Behavioral Patterns and Communication and Interaction).
Toilet Training | for 8 weeks, once a week
  It was developed to assess mothers' knowledge and attitudes towards toilet training. The scale consists of 29 Likert-type items, ranging from 1 to 5 (5-Strongly Agree, 4-Agree, 3-Don't Know, 2-Disagree, 1-Strongly Disagree), which measure mothers' preferences for agreeing or disagreeing with toilet training 25 knowledge and attitudes. The scale does not contain reverse items or scoring. A minimum of 1 and a maximum of 5 points can be obtained from the scale items. As the scale score increases, mothers' knowledge and attitudes towards Toilet Training increase positively.
Readiness to Stop Breastfeeding | for 8 weeks, once a week
  It is a 5-point Likert-type scale (1 = Strongly Disagree, 2 = Disagree, 3 = Somewhat Agree, 4 = Agree, 5 = Strongly Agree). It can be applied to all mothers with babies 18 months and older. Items 2, 5, 13, 15, and 16 on the scale need to be reverse coded. The total score that can be obtained from the scale varies between 19-95. As the scores obtained from the scale increase, it is interpreted that the level of Readiness to Stop Breastfeeding increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Iğdır University, Iğdır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No